CLINICAL TRIAL: NCT01742871
Title: Nutritional Status of Patients Victims of Haemorragic Accidents With Antivitamins K
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0131; 2012-A00331-42
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hemorrhagic Accident; Iatrogeny; Denutrition
Keywords: Antivitamin K; Bleeding; Haemorrhage; Nutritional status; impedancemetry
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- controls: Patient under anti-vitamin K with no haemorrhagic manifestations admitted for another reason to Emergency Adults
- kaskadil: Patient under anti-vitamin K with a serious bleeding event that required treatment in the emergency Adults. Is considered serious accident requiring the use of a reversion by PPSB (Kaskadil ®).

SUMMARY:
Bleeding under vitamin K antagonists are a major iatrogenic causes of hospitalization, subject to a fatal outcome in more than one third of cases, mortality is particularly high in cases of serious bleeding, including intracerebral hemorrhage. If the INR measured in these patients are often away from the higher value of the target range, a significant proportion of bleeding were observed for INR between 2 and 3. The study captures the components of the nutritional status of patients on oral anticoagulants, including any micronutrient deficiencies, to determine whether nutritional status is an independent risk factor for bleeding

DETAILED DESCRIPTION:
Be included in this study patients under anti-vitamin K supported or followed the emergency department Adults.

The inclusion visit will be conducted in the emergency department Adults Clermont-Ferrand by an emergency physician or investigator or co-investigator. The protocol will be explained to patients in detail, the information document and consent will be issued for playback, then they will be asked to sign the consent form and participation agreement.

Case-control study: patients under oral anticoagulant with severe hemorrhagic accident compared with patients without hemorrhagic accident. Cases will be matched to controls based on age, sex, and the value of the INR.

Patients will be divided into two groups:

* Group 1: cases Patient under anti-vitamin K with a serious bleeding event that required treatment in the emergency Adults. Is considered serious accident requiring the use of a reversion by PPSB (Kaskadil ®).
* Group 2: contols Patient under anti-vitamin K with no haemorrhagic manifestations admitted for another reason to Emergency Adults

Each case will be paired with two controls

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, aged over 18, under oral anticoagulant therapy with antivitamins K.
* INR greater than 1.5, in the therapeutic range or overdose
* Patient have read, understood and signed the consent form or inclusion emergency consent of the person with confidence
* Case-control study: patients under oral anticoagulant with severe hemorrhagic accident compared with patients without hemorrhagic accident. Cases will be matched to controls based on age, sex, and the value of INR :

Case:

Patients victims of serious hemorrhagic accident on VKAs, supported emergency Adults.

Will be considered severe hemorrhagic stroke, accidents requiring the use of a reversion by PPSB (Kaskadil ®)

Control :

Patients on VKAs supported the Emergency Adults for a reason other than bleeding.

Exclusion Criteria:

* underage patients
* Patients who have not read or understood nor signed the consent form or refusal of the reference person.
* pregnant women
* Patients with a pacemaker and / or implantable defibrillator
* Patients with mechanical valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Be included in this study patients under anti-vitamin K supported or followed the emergency department Adults.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Denutrition diagnosis | at day 1

SECONDARY OUTCOMES:
Zinc blood level | at day 1
Cupper blood level | at day 1
vitamin C blood level | at day 1
vitamin B1 blood level | at day 1
PINI (pronostic inflammatory and nutritional index) | at day 1
NRI (nutritional risk index) | at day 1
The outpatient bleeding risk index | at day 1
Stiffness index | at day 1
Rumpel-Leede test | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moustafa F, Dopeux L, Mulliez A, Boirie Y, Morand C, Gentes E, Farigon N, Richard D, Lebreton A, Teissandier D, Dutheil F, Schmidt J. Severe undernutrition increases bleeding risk on vitamin-K antagonists. Clin Nutr. 2021 Apr;40(4):2237-2243. doi: 10.1016/j.clnu.2020.10.002. Epub 2020 Oct 9. PMID 33077273